CLINICAL TRIAL: NCT06012149
Title: Braining: Implementation of Physical Exercise for Patients in Specialist Psychiatry, Efficacy Evaluation in a Randomized Controlled Multicentre Trial
Brief Title: Braining: Implementation of Physical Exercise for Patients in Specialist Psychiatry
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-07130
Record Dates: First submitted 2023-07-07; First posted 2023-08-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mental Disorders
Keywords: physical exercise; mental disorders
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled superiority trial evaluating if the new method Braining is superior to structured advice on physical activity, concerning increasing physical activity.
  The trial is a multicenter study conducted at 3-6 sites. Participants are individually randomized in blocks of 2-4 at each site.
Who Masked: Investigator
Masking Description: Intervention will be blinded to investigators during analysis of primary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braining (Experimental): A 12 week program where participants are encouraged to participate in physical exercise at the psychiatric unit.
  Interventions: Behavioral: Braining
- Structured advice on physical activity (Active Comparator): Health interview and a 12 week program where participants are encouraged to engage in physical exercise outside the psychiatric setting.
  Interventions: Behavioral: Structured advice on physical activity

INTERVENTIONS:
Behavioral: Braining — A 12 week program where participants are encouraged to participate in physical exercise at the psychiatric unit.
  Arms: Braining
Behavioral: Structured advice on physical activity — A 12 week program where participants are encouraged to engage in physical exercise
  Other Names: Advice on physical activity
  Arms: Structured advice on physical activity

SUMMARY:
The goal of this clinical trial is to compare Braining, a physical exercise lifestyle intervention in psychiatric care, with structured advice on physical exercise.

The main questions are:

* does Braining lead to increased physical exercise compared to structured advice on physical exercise?
* what effect does Braining have on mental and physical health, quality of life and functional level compared to structured advice on physical exercise?

The participants will join a twelve weeks long study period with clinician led exercise classes up to three times per week. Before and after the study period they will leave blood tests, take part in a mental and physical examination and fill in assessment scales. To measure physical activity, the participants will carry an accelerometer, a device that measures steps and acceleration. After six and twelve months, the participants take part in the same measurements.

The control group takes parts in the same measurements and follow up, but instead of having clinician led exercise classes, they will exercise on their own during the twelve weeks study period.

DETAILED DESCRIPTION:
Braining is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic moderate to vigorous aerobic group training sessions and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan. Braining is unique in that it:

1. Includes trained psychiatric clinical staff exercising together with patients from both out- and inpatient ward units in daily, moderate to vigorous aerobic group training sessions
2. is included in regular healthcare fee, (free of charge)
3. includes a motivational and educational visit (as a group seminar or as an individual visit) at the start and end of a twelve-week exercise intervention
4. includes regular measurements (self-assessment questionnaires, blood samples, physical and mental health examination and education before and after the twelve-week exercise intervention)
5. offers short individual motivating visits before every training session, including assessment of day shape and fitness to participate.

This study will be a multi-center study performed at 5 psychiatric outpatient units in Region Stockholm. Patients with symptoms of depression and/or anxiety who are not physically active in accordance with WHO recommendations will be invited to participate in the study.

The research questions are:

* Does Braining increase the amount of completed physical training (PT) compared to structured advice on physical exercise (advice on PT according to guidelines)?
* What effect does Braining have on the mental and physical health, quality of life and functional level of participating patients compared to structured advice on physical exercise? Examined from the following points of view:

  * psychiatric symptoms, such as depression, anxiety, insomnia, emotional regulation?
  * somatic symptoms, such as blood pressure, resting heart rate, BMI, waist measurement, presence of somatic co-morbidity?
* How do participants rate Braining and structured advice on physical exercise regarding:

  1. Satisfaction with treatment
  2. Credibility of treatment
  3. Negative effects
* Is Braining a cost-effective intervention?

Participants will be randomized to supplementary treatment with Braining or structured advice on physical activity.

Braining and advice on physical activity will be compared after a 12-week training period.

Measurements of the participants´ psychiatric and somatic health are carried out before the treatment, after 4, 8 and 12 weeks and 6 and 12 months after the end of treatment. Effects of the treatment are examined via validated self-assessment forms, as well as somatic examination with a focus on metabolic status. Venous blood samples are taken before and after the 12-week training period, as well as 6 and 12 months after the end of the training period to investigate changes in metabolic status. In a sub study on a smaller number of participants the researchers will analyze associations with biological factors such as genetic or epigenetic factors, metabolic factors, stress hormone levels, trace elements, degree of inflammation and other biological markers of health and disease that can be measured in ordinary blood tests, e.g. through "Omik" design. Physical activity will be measured by self assessment scales, accelerometer and by number of performed Braining classes.

Data analysis plan Continuous data will be analyzed using mixed effects models. The interaction effect of group and time will be the central estimate of the effect of the intervention Braining.

The primary analyses will follow the intention-to-treat principle and include all randomized participants. Adjusted as well as unadjusted results from analyses will be reported. Analyses will be adjusted for prespecified covariates to improve precision. Covariates adjusted for in the primary and secondary analysis will be age, sex, and unit where participants were registered as patients.

Missing data will be handled with multiple imputation with chained equations (MICE) to minimize bias compared to listwise deletion or single imputation and reflect the uncertainty caused by missingness. For each outcome, 20 datasets will be imputed and analyzed, pooling the results.

Per protocol analyses will be conducted as sensitivity analyses, including participants with at least 75% adherence to the intervention, defined as completion of ≥3 of 4 scheduled intervention visits. In the Braining arm, additional adherence will be defined as completion of at least eight Braining sessions. This approach is intended to estimate the effect of the intervention under conditions of adequate adherence.

Sensitivity analyses will examine the impact of alternative ActivPAL data validity criteria by restricting the sample to participants with 4-7 valid days of ActivPAL data. This analysis is intended to evaluate the robustness of the results to different assumptions regarding accelerometer data completeness.

Subgroup analysis:

* Will explore whether continuous variables of baseline depression severity, according to PHQ-9, moderate treatment effects in PHQ-9 and ActivPAL/MVPA.
* Will explore whether continuous variables of baseline physical activity levels, according to ActivPAL/MVPA, moderate treatment effects in primary analysis in ActivPAL/MVPA and PHQ-9.
* Will be conducted among participants with metabolic syndrome, defined as the presence of three or more cardiometabolic risk factors.

These analyses are considered secondary/exploratory and will be interpreted cautiously.

ELIGIBILITY:
Inclusion Criteria:

* Patient at one of the psychiatric units

Exclusion Criteria:

* Physically active with moderate to vigorous physical activity above recommendations from World Health Organization (WHO) during the last 4 weeks
* Severe mental disorder such as ongoing mania, psychosis, and conditions when high risk of suicide or high risk of violence available according to the assessment of psychiatric staff at the unit.
* Medical conditions such as heart or lung disease, infection, withdrawal, where heart rate-increasing physical activity is considered contraindicated due to Medical reasons.
* Physical disability that makes it impossible to move independently to the gym and performing the indicated exercise in the training sessions.
* Mental disability which means that you can not participate in group training.
* Difficulty speaking or understanding the Swedish language.
* Ongoing heavy substance use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Change from Pre intervention start to 12 weeks post intervention start
  Moderate to vigorous intensity physical activity (MVPA) objectively measured with the ActivPAL accelerometer, operationalized as >100 steps per minute (SPM) and potentially vigorous intensity physical activity (VPA) > 125 SPM with ActivPAL.
Patient Health Questionnaire 9 (PHQ-9) | Change from Pre intervention start to 12 weeks post intervention start
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.

SECONDARY OUTCOMES:
Physical activity | Change from Pre intervention start to 6 months post intervention start
  Moderate to vigorous intensity physical activity (MVPA) objectively measured with the ActivPAL accelerometer, operationalized as >100 Steps per minute (SPM) and potentially vigorous intensity physical activity (VPA) > 125 SPM with ActivPAL.
Physical activity | Change from Pre intervention start to 12 months post intervention start
  Moderate to vigorous intensity physical activity (MVPA) objectively measured with the ActivPAL accelerometer, operationalized as >100 Steps per minute (SPM) and potentially vigorous intensity physical activity (VPA) > 125 SPM with ActivPAL.
Self reported physical activity | Change from Pre intervention start to 12 weeks post intervention start
  Self-reported physical activity: Total physical activity as Metabolic Energy Turnover (MET)hours/week and three level categories (low, moderate and high).
Self reported physical activity | Change from Pre intervention start to 6 months post intervention start
  Self-reported physical activity: Total physical activity as Metabolic Energy Turnover (MET)hours/week and three level categories (low, moderate and high).
Self reported physical activity | Change from Pre intervention start to 12 months post intervention start
  Self-reported physical activity: Total physical activity as Metabolic Energy Turnover (MET)hours/week and three level categories (low, moderate and high).
Patient Health Questionnaire 9 (PHQ-9) | Change from Pre intervention start to 6 months post intervention start
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
Patient Health Questionnaire 9 (PHQ-9) | Change from Pre intervention start to 12 months post intervention start
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Change from Pre intervention start to 12 weeks post intervention start
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Change from Pre intervention start to 6 months post intervention start
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Change from Pre intervention start to 12 months post intervention start
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Insomnia Severity Index (ISI) | Change from Pre intervention start to 12 weeks post intervention start
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
Insomnia Severity Index (ISI) | Change from Pre intervention start to 6 months post intervention start
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
Insomnia Severity Index (ISI) | Change from Pre intervention start to 12 months post intervention start
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
The Work and Social Adjustment Scale (WSAS) | Change from Pre intervention start to 12 weeks post intervention start
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from Pre intervention start to 6 months post intervention start
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from Pre intervention start to 12 months post intervention start
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better. The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
EUROQOL 5 dimensions (EQ5D) | Change from Pre intervention start to 12 weeks post intervention start
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
EUROQOL 5 dimensions (EQ5D) | Change from Pre intervention start to 6 months post intervention start
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
EUROQOL 5 dimensions (EQ5D) | Change from Pre intervention start to 12 months post intervention start
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
Quality Adjusted Life Years (QALY) | Change from 12-0 months pre intervention to 0-12 months post intervention
  The quality-adjusted life year (QALY) is a generic measure of disease burden, including both the quality and the quantity of life lived. It is used in economic evaluation to assess the value of medical interventions. One QALY equates to one year in perfect health. QALY scores range from 1 (perfect health) to 0 (dead).
The incremental cost-effectiveness (ICER) | Change from 12-0 months pre intervention to 0-12 months post intervention
  The incremental cost-effectiveness ratio (ICER) is a statistic used in cost-effectiveness analysis to summarise the cost-effectiveness of a health care intervention. It is defined by the difference in cost between two possible interventions, divided by the difference in their effect. It represents the average incremental cost associated with 1 additional unit of the measure of effect. Costs will be described in monetary units, while effects will be measured in terms of health status.
Blood pressure | Change from Pre intervention start to 12 weeks post intervention start
  systolic and diastolic, mmHg
Blood pressure | Change from Pre intervention start to 6 months post intervention start
  systolic and diastolic, mmHg
Blood pressure | Change from Pre intervention start to 12 months post intervention start
  systolic and diastolic, mmHg
Body mass index (BMI) | Change from Pre intervention start to 12 weeks post intervention start
  Weight in kg divided by the square of height in m
Body mass index (BMI) | Change from Pre intervention start to 6 months post intervention start
  Weight in kg divided by the square of height in m
Body mass index (BMI) | Change from Pre intervention start to 12 months post intervention start
  Weight in kg divided by the square of height in m
Waist circumference | Change from Pre intervention start to 12 weeks post intervention start
  Waist circumference, cm
Waist circumference | Change from Pre intervention start to 6 months post intervention start
  Waist circumference, cm
Waist circumference | Change from Pre intervention start to 12 months post intervention start
  Waist circumference, cm
Heart rate (HR) | Change from Pre intervention start to 12 weeks post intervention start
  Heart rate, beats per minute, resting state
Heart rate (HR) | Change from Pre intervention start to 6 months post intervention start
  Heart rate, beats per minute, resting state
Heart rate (HR) | Change from Pre intervention start to 12 months post intervention start
  Heart rate, beats per minute, resting state
fasting blood sugar (FBS) | Change from Pre intervention start to 12 weeks post intervention start
  fasting blood sugar, mmol/l
fasting blood sugar (FBS) | Change from Pre intervention start to 6 months post intervention start
  fasting blood sugar, mmol/l
fasting blood sugar (FBS) | Change from Pre intervention start to 12 months post intervention start
  fasting blood sugar, mmol/l
Hemoglobin A1c (HbA1c) | Change from Pre intervention start to 12 weeks post intervention start
  Glycated hemoglobin, mmol/mol
Hemoglobin A1c (HbA1c) | Change from Pre intervention start to 6 months post intervention start
  Glycated hemoglobin, mmol/mol
Hemoglobin A1c (HbA1c) | Change from Pre intervention start to 12 months post intervention start
  Glycated hemoglobin, mmol/mol
Blood lipids | Change from Pre intervention start to 12 weeks post intervention start
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | Change from Pre intervention start to 6 months post intervention start
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | Change from Pre intervention start to 12 months post intervention start
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Sensitive C-reactive protein (CRP) | Change from Pre intervention start to 12 weeks post intervention start
  Measurement of inflammation and infection, mmol/L
Sensitive C-reactive protein (CRP) | Change from Pre intervention start to 6 months post intervention start
  Measurement of inflammation and infection, mmol/L
Sensitive C-reactive protein (CRP) | Change from Pre intervention start to 12 months post intervention start
  Measurement of inflammation and infection, mmol/L
Complete blood count | Change from Pre intervention start to 12 weeks post intervention start
  The number of leukocytes, platelets and erythrocytes per unit volume in a sample of venous blood. Includes measurement of the hemoglobin, hematocrit and erythrocyte indices.
Complete blood count | Change from Pre intervention start to 6 months post intervention start
  The number of leukocytes, platelets and erythrocytes per unit volume in a sample of venous blood. Includes measurement of the hemoglobin, hematocrit and erythrocyte indices.
Complete blood count | Change from Pre intervention start to 12 months post intervention start
  The number of leukocytes, platelets and erythrocytes per unit volume in a sample of venous blood. Includes measurement of the hemoglobin, hematocrit and erythrocyte indices.
Negative effects | 12 weeks post inclusion
  Self constructed question regarding if participants have had any negative effects of treatment: 1) Have you experienced any negative effects from the treatment 2) If yes, please specify:
The Client Satisfaction Questionnaire-8 (CSQ-8) | 12 weeks post inclusion
  Self rated satisfaction of treatment. Minimum value 8, maximum value 32 where higher values indicate greater satisfaction with the treatment.
The Credibility/Expectancy Questionnaire (CEQ) | 2 weeks post inclusion
  Self rated Credibility of treatment. Minimum value 3, maximum value 27 for each factor, where higher values indicate greater Credibility/Expectancy of the treatment.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from Pre intervention start to 12 weeks post intervention start
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from Pre intervention start to 6 months post intervention start
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale, Brief Version (DERS-16) | Change from Pre intervention start to 12 months post intervention start
  Self rated difficulties in emotion regulation. The sum ranges from 16 to 80, where higher levels indicate greater difficulty in emotion regulation.
Time Line follow back (TLFB) | Change from Pre intervention start to 12 weeks post intervention start.
  Interview regarding alcohol and/or drug intake, measuring number of days with alcohol/drug consumption.
Time Line follow back (TLFB) | Change from Pre intervention start to 6 months post intervention start.
  Interview regarding alcohol and/or drug intake, measuring number of days with alcohol/drug consumption.
Time Line follow back (TLFB) | Change from Pre intervention start to 12 months post intervention start.
  Interview regarding alcohol and/or drug intake, measuring number of days with alcohol/drug consumption.
The Alcohol Use Disorders Identification Test (Audit - C) | Change from Pre intervention start to 12 weeks post intervention start.
  AUDIT-C is an alcohol screen that can help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
The Alcohol Use Disorders Identification Test (Audit - C) | Change from Pre intervention start to 6 months post intervention start.
  AUDIT-C is an alcohol screen that can help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
The Alcohol Use Disorders Identification Test (Audit - C) | Change from Pre intervention start to 12 months post intervention start.
  AUDIT-C is an alcohol screen that can help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Physical Activity | Change from Pre intervention start to 12 weeks post intervention start
  Sit to stand transitions, steps per day, sedentary time, and time in light intensity physical activity measured with the ActivPAL accelerometer.
Physical Activity | Change from Pre intervention start to 6 months post intervention start.
  Sit to stand transitions, steps per day, sedentary time, and time in light intensity physical activity measured with the ActivPAL accelerometer.
Physical activity | Change from pre intervention start to 12 months past intervention start.
  Sit to stand transitions, steps per day, sedentary time, and time in light intensity physical activity measured with the ActivPAL accelerometer.

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Region Stockholm, Psykiatri Sydväst (Psychiatric Clinic Psychiatry Southwest), Stockholm, Stockholm County
  - Region Stockholm, Psykiatri Nordväst och Beroendecentrum, mottagningar Väsby, Upplands Vasby, Stockholm County
  - Region Stockholm, Beroendecentrum, Magnus Huss, Stockholm
  - Region Stockholm, Liljeholmsberget, Stockholm
  - Region Stockholm, Psykiatri Södra, Andreashuset, Stockholm

IPD SHARING:
Plan to Share IPD: No